CLINICAL TRIAL: NCT00527124
Title: A Randomized, Phase II Trial of AZD2171, Docetaxel, and Prednisone Compared to Docetaxel and Prednisone in Patients With Metastatic, Hormone Refractory Prostate Cancer
Brief Title: Docetaxel and Prednisone With or Without Cediranib in Treating Patients With Metastatic Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Closure was recommended by CTEP due to slow accrual.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00174; NCI-2009-00174 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007-015 (Other: Barbara Ann Karmanos Cancer Institute); CDR0000564449 (Registry Identifier: Clinicaltrials.gov); 2007-015 (Other: Wayne State University); 7451 (Other: CTEP); N01CM00038 (NIH); U01CA062491 (NIH); P30CA022453 (NIH); U01CA062487 (NIH)
Record Dates: First submitted 2007-09-07; First posted 2007-09-10 (Estimated); Results first posted 2014-03-11 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-07

CONDITIONS: Adenocarcinoma of the Prostate; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cediranib; Docetaxel; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral cediranib maleate once daily on days 1-21, docetaxel IV over 1 hour on day 1, and oral prednisone twice daily on days 1-21.
  Interventions: Drug: cediranib maleate; Drug: docetaxel; Drug: prednisone; Other: laboratory biomarker analysis
- Arm II (Active Comparator): Patients receive docetaxel and prednisone as in arm I.
  Interventions: Drug: docetaxel; Drug: prednisone; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
  Arms: Arm I
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Drug: prednisone — Given orally
  Other Names: DeCortin; Deltra
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well giving docetaxel and prednisone together with or without cediranib works in treating patients with metastatic prostate cancer that did not respond to hormone therapy. Drugs used in chemotherapy, such as docetaxel and prednisone, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Cediranib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Giving docetaxel together with prednisone, with or without cediranib, may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 6-month progression-free survival rate of patients with hormone refractory metastatic adenocarcinoma of the prostate treated with docetaxel and prednisone with vs without cediranib.

SECONDARY OBJECTIVES:

I. To evaluate the safety profile of cediranib, docetaxel, and prednisone in patients with metastatic hormone-refractory prostate cancer.

II. To determine the duration of prostate-specific antigen (PSA) response and PSA control in patients with metastatic hormone-refractory prostate cancer treated with cediranib, docetaxel, and prednisone.

III. To determine the partial and complete response rate in patients with measurable disease treated with cediranib, docetaxel, and prednisone.

IV. To determine time to progression in patients with metastatic hormone-refractory prostate cancer treated with cediranib, docetaxel, and prednisone.

V. To determine overall survival in patients with metastatic hormone-refractory prostate cancer.

VI. To perform correlative marker studies measuring serum levels of VEGF, PDGF, sICAM, bFGF, interleukin (IL)-6, and IL-8.

VII. To perform a pilot study of [F18]FMAU positron emission test (PET) imaging on patients receiving cediranib, docetaxel, and prednisone.

OUTLINE: This is a multicenter study. Patients are stratified by participating institution. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral cediranib once daily on days 1-21, docetaxel IV over 1 hour on day 1, and oral prednisone twice daily on days 1-21.

ARM II: Patients receive docetaxel and prednisone as in arm I.

In both arms, courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. Archival paraffin-embedded tissue blocks or slides from time of diagnosis (or subsequent, but prior to therapy) are evaluated for expression of molecular targets relevant to this study. Blood specimens from baseline, after courses 1 and 2, and after completion of study treatment are analyzed for protein markers. Samples are analyzed by ELISA and IHC for angiogenesis-associated plasma proteins, plasma levels of VEGF, tumor expression of PDGFR, and interleukin (IL)-6 and IL-8 plasma levels. Patients also undergo positron emission test (PET) scans utilizing fluorodeoxyglucose (FDG) at baseline and after course 1.

After completion of study treatment, patients are followed every 3 months for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Clinical/radiologic metastases with objective evidence of disease progression by imaging or by rising prostate-specific antigen (PSA) despite androgen deprivation therapy
* Rising PSA must be determined based on a rising trend with 2 successive elevations at a minimum interval of 1 week
* Meets 1 of the following criteria: Measurable disease, with any level of PSA, at least 1 unidimensionally measurable lesion (longest diameter to be recorded) >= 20 mm by conventional techniques or >= 10 mm by spiral CT scan, nonmeasurable disease, PSA >= 5 ng/mL OR new areas of bony metastases on bone scan
* Castrate levels of testosterone < 50 ng/dL must be maintained and documented
* Luteinizing hormone-releasing hormone (LHRH) agonist therapy must be continued, if required to maintain castrate levels of testosterone
* Total bilirubin normal
* Patients with radiological evidence of stable brain metastases are eligible provided they are asymptomatic and do not require corticosteroids or have been treated with corticosteroids and show clinical and radiological evidence of stabilization at least 10 days after discontinuation of steroids
* ECOG performance status (PS) =< 2 or Karnofsky PS 60-100%
* Life expectancy > 12 weeks
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelet count >= 100,000/mcL
* Histologically confirmed adenocarcinoma of the prostate
* AST and ALT =< 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Proteinuria =< 1+ and urine protein:creatinine ratio =< 1.0 OR 24-hour urine protein < 1,000 mg
* Peripheral neuropathy >= grade 2
* Uncontrolled intercurrent illness including, but not limited to, any of the following: ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, psychiatric illness/social situations that would limit compliance with study requirements
* Congestive heart failure, second or third degree heart block, or recent myocardial infarction within the past 6 months
* QTc prolongation > 500 msec OR other ECG abnormality noted within 14 days of treatment
* New York Heart Association class III or IV cardiac disease; Class II disease controlled with treatment and monitoring allowed
* History of poorly controlled hypertension (e.g., resting blood pressure > 150/90 mm Hg with or without hypertensive therapy)
* History of a curatively treated malignancy with a survival prognosis of less than 5 years or concurrent malignancy except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ
* History of significant gastrointestinal impairment, as judged by the investigator, that would significantly affect the absorption of cediranib
* History of severe hypersensitivity reaction to docetaxel or other drugs formulated with polysorbate 80
* Significant hemorrhage (30 mL bleeding/episode in previous 3 months) or hemoptysis (5 mL fresh blood in previous 4 weeks)
* Prior enrollment or randomization of treatment in the present study
* Patients must be off flutamide antiandrogen therapy for ≥ 4 weeks (6 weeks for bicalutamide or nilutamide)
* No prior chemotherapy for metastatic prostate cancer
* No major surgery within the past 14 days or a surgical incision that is not fully healed
* No HIV-positive patients on combination antiretroviral therapy
* No conditions requiring concurrent use of drugs or biologics with proarrhythmic potential
* No other investigational agents within 30 days prior to study enrollment
* No untreated unstable brain or meningeal metastases
* Known hypersensitivity to cediranib or any of its excipients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2007-11; Primary Completion 2012-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Heath, Principal Investigator — Wayne State University
Locations (4):
- United States (4):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Wayne State University, Detroit, Michigan
  - M D Anderson Cancer Center, Houston, Texas
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from the outpatient clinics or inpatient service of Karmanos Cancer Center by physicians in the Department of Hematology and Medical Oncology, between December 2007 and December 2011.
Pre-assignment Details: 57 subjects went on study; an additional 27 subjects were consented, 23 were not eligible to go on study, 4 withdrew from study.
Groups:
- Arm I: Patients receive oral cediranib once daily on days 1-21, docetaxel IV over 1 hour on day 1, and oral prednisone twice daily on days 1-21.
Period: Overall Study
Arm/Group | Arm I | Arm II
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.14 (7.3) | 68.29 (9.66) | 68.72 (8.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 29 | 28 | 57
Region of Enrollment [Number; unit: participants]
  United States | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: 6-month Progression-free Survival (PFS) Proportion
Description: The proportion of patients on each treatment arm who survive ≥ 6.00 months progression-free
Time Frame: Followed for 52 weeks at 3 month intervals after coming off treatment, time period equal to the length of treatment + up to 12 months
Population: Per protocol. 30 subjects on Arm I and 28 subjects on Arm II accrued for analysis of the primary endpoint of 6 mths PFS proportion. PFS is obtainable on all 58 participants enrolled, however 1 subject enrolled on Arm I withdrew before receiving any treatment, hence cannot be included for AE analysis and reporting, AE results involve 29 subjects.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Groups:
- Arm I: Patients receive oral cediranib 20 mg once daily on days 1-21, docetaxel 75mg/m2 IV over 1 hour on day 1 every 3 weeks, and oral prednisone 5mg twice daily on days 1-21.
- Arm II: Patients receive docetaxel 75 mg/m2 IV every 3 weeks, and prednisone 5mg orally twice a day, Repeat cycle every 21 days.
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 30 | 28
percentage of patients | 60 [42 to 75] | 54 [36 to 71]
Statistical Analysis 1: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.7428, Regression, Cox; Hazard Ratio (HR) = 0.907, 95% CI 2-sided [0.506 to 1.624], Standard Error of Mean 0.29730
Statistical Analysis 2: Comparison: Arm I vs Arm II; Test type: Superiority or Other; p = 0.7425, Log Rank

2. Secondary Outcome: Prostate-specific Antigen (PSA) Response in Accordance With the Prostate Specific Antigen Working Group
Description: PSA < 4.0 ng/ml. is a CR. A 50% decline or better in PSA is a PR. Less than a 50% decline in PSA and less than a 25% increase in PSA is SD. A 25% or greater increase in PSA level by at least 5 ng/mL is PD by PSA only. The point estimate and 95% Wilson CI estimates of the proportion for the Prostate-specific antigen (PSA) response will be computed .
Time Frame: Up to 52 weeks
Measure: Number (95% Confidence Interval); unit: proportion of evaluable patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 30 | 28
proportion of evaluable patients
  CR | .35 [.19 to .54] | .12 [.04 to .29]
  PR | .27 [.14 to .46] | .54 [.35 to .71]
  SD | .35 [.19 to .54] | .31 [.17 to .50]
  PD | .04 [.01 to .19] | .04 [.01 to .19]

3. Secondary Outcome: Overall Response Rate Evaluated by the RECIST Criteria
Description: The overall response is determined by combining the patient's status on target lesions, PSA, non-target lesions, and new disease as defined in the following table.
  Target Lesions CR CR PR SD PD Any Any Any
  PSA Response CR PR PR Non-PD Any Any PD Any
  Non-Target Lesions CR Non-CR/Non-PD Non-PD Non-PD Any PD Any Any
  New Lesions No No No No Yes or No Yes or No Yes or No Yes
  Overall Response CR PR PR SD PD PD PD PD
Time Frame: Up to 52 weeks
Measure: Number (95% Confidence Interval); unit: proportion of evaluable patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 30 | 28
proportion of evaluable patients
  SD | .92 [.75 to .98] | .92 [.76 to .98]
  PD | .08 [.02 to .25] | .08 [.02 to .24]

4. Secondary Outcome: Time to Progression
Description: Analyzed with standard K-M methodology. Both point and 95% CI estimates of the median and other statistics (e.g., the 3-month rate, 6-month rate, etc.) will be computed from the censored distribution of TTP. These point and CI estimates will be reported for all patients combined, and separately for each treatment arm.
Time Frame: The time from registration date until documented clinical disease progression, or until date of death, whichever occurs first, assessed up to 52 weeks
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 30 | 28
months | 8.0 [4.2 to 11.9] | 6.4 [4.8 to 10.2]

5. Secondary Outcome: Overall Survival
Description: Analyzed with standard K-M methodology. A 12 month survival rate will be calculated since median survival was not reached by the end of the study period.
Time Frame: The time from registration date until death from any cause, assessed up to 52 weeks
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Arm I | Arm II
Number analyzed (Participants) | 30 | 28
percentage of patients | 71 [51 to 84] | 76 [55 to 88]

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II
Serious Adverse Events (participants affected / at risk) | 20/29 | 9/28
Other Adverse Events (participants affected / at risk) | 29 | 28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=29) | Arm II (N=28)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Febrile netropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiopulmonary arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Chest pain-cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Rectal hemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Infection with Grade 3 or 4 Neutrophils (ANC <1.0 X 10E9/L): Bronchus (Infections and infestations) | 0 (0) | 1 (1)
Infection with Grade 3 or 4 Neutrophils (ANC <1.0 X 10E9/L): Lung (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 5 (5) | 1 (1)
Neutrophil count decreased (Investigations) | 12 (12) | 3 (3)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 11 (11) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Ischemia cerebrovascular (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 5 (5) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 3 (3) | 0 (0)
Thromboembolic event (Vascular disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Arm I | Arm II
Anemia (Blood and lymphatic system disorders) | 16/29 (16) | 16/28 (16)
Chest pain- cardiac (Cardiac disorders) | 0/29 (0) | 2/28 (2)
Watering eyes (Eye disorders) | 5/29 (5) | 3/28 (3)
Abdominal pain (Gastrointestinal disorders) | 4/29 (4) | 0/28 (0)
Diarrhea (Gastrointestinal disorders) | 6/29 (6) | 25/28 (25)
Dyspepsia (Gastrointestinal disorders) | 2/29 (2) | 3/28 (3)
Mucositis oral (Gastrointestinal disorders) | 2/29 (2) | 10/28 (10)
Rectal hemorrhage (Gastrointestinal disorders) | 0/29 (0) | 2/28 (2)
Vomiting (Gastrointestinal disorders) | 2/29 (2) | 6/28 (6)
Edema limbs (General disorders) | 8/29 (8) | 5/28 (5)
Fatigue (General disorders) | 15/29 (15) | 23/28 (23)
Fever (Gastrointestinal disorders) | 2/29 (2) | 0/28 (0)
Urinary tract infection (Infections and infestations) | 2/29 (2) | 2/28 (2)
Alanine aminotransferase increased (Investigations) | 4/29 (4) | 9/28 (9)
Creatinine increased (Investigations) | 4/29 (4) | 5/28 (5)
INR increased (Investigations) | 0/29 (0) | 2/28 (2)
Lymphocyte count decreased (Investigations) | 13/29 (13) | 16/28 (16)
Neutrophil count decreased (Investigations) | 13/29 (13) | 9/28 (9)
Platelet count decreased (Investigations) | 8/29 (8) | 15/28 (15)
White blood cell decreased (Investigations) | 11/29 (11) | 11/28 (11)
Anorexia (Metabolism and nutrition disorders) | 5/29 (5) | 12/28 (12)
Dehydration (Metabolism and nutrition disorders) | 0/29 (0) | 4/28 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 12/29 (12) | 15/28 (15)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13/29 (13) | 15/28 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 6/29 (6) | 13/28 (13)
Hypoglycemia (Metabolism and nutrition disorders) | 3/29 (3) | 3/28 (3)
Hyponatremia (Metabolism and nutrition disorders) | 5/29 (5) | 11/28 (11)
Hypophosphatemia (Metabolism and nutrition disorders) | 5/29 (5) | 6/28 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 3/29 (3) | 5/28 (5)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3/29 (3) | 2/28 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 2/29 (2) | 0/28 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4/29 (4) | 7/28 (7)
Proteinuria (Renal and urinary disorders) | 2/29 (2) | 11/28 (11)
Urinary incontinence (Renal and urinary disorders) | 0/29 (0) | 2/28 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4/29 (4) | 10/28 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2/29 (2) | 10/28 (10)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0/29 (0) | 10/28 (10)
Rash acneiform (Skin and subcutaneous tissue disorders) | 0/29 (0) | 2/28 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0/29 (0) | 4/28 (4)
Hypotension (Vascular disorders) | 0/29 (0) | 3/28 (3)

LIMITATIONS AND CAVEATS:
Closure was recommended by CTEP due to slow accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less